CLINICAL TRIAL: NCT03539601
Title: A PHASE 3B/4, MULTICENTER, RANDOMIZED, ASSESSOR BLINDED, VEHICLE AND ACTIVE (TOPICAL CORTICOSTEROID AND CALCINEURIN INHIBITOR) CONTROLLED, PARALLEL GROUP STUDY OF THE EFFICACY, SAFETY, AND LOCAL TOLERABILITY OF CRISABOROLE OINTMENT, 2% IN PEDIATRIC AND ADULT SUBJECTS (AGES 2 YEARS AND OLDER) WITH MILD TO MODERATE ATOPIC DERMATITIS
Brief Title: A Study of Crisaborole Ointment 2%; Crisaborole Vehicle; TCS and TCI in Subjects Aged ≥ 2 Years, With Mild-moderate AD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This decision was made for business reasons only and is not related to any safety concerns regarding crisaborole.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C3291037; 2018-001043-31 (EudraCT Number)
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Results first posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis, Crisaborole ointment 2%, TCS, TCI
MeSH Terms: conditions — Dermatitis, Atopic; Mandibulofacial Dysostosis | interventions — crisaborole; pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigational products above are masked for appearance, and will be placed into identical cartons. Once removed from the product cartons, the investigational products could be discerned from each other based on commercial product tube shape/size and should only be handled by unblinded site personnel.
  Safety and efficacy assessments will be conducted at the investigator site by a clinical assessor blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Crisaborole ointment, 2% (Experimental): This treatment arm will be administered both in Cohort 1 and Cohort 2.
  Interventions: Drug: Crisaborole ointment, 2%
- Hydrocortisone butyrate cream, 0.1% (Active Comparator): This treatment arm will be administered in Cohort 1 only.
  Interventions: Drug: Hydrocortisone butyrate cream, 0.1%
- Pimecrolimus cream, 1% (Active Comparator): This treatment arm will be administered in Cohort 2 only.
  Interventions: Drug: Pimecrolimus cream, 1%
- Crisaborole Vehicle (Placebo Comparator): This treatment arm will be administered both in Cohort 1 and Cohort 2.
  Interventions: Drug: Crisaborole Vehicle

INTERVENTIONS:
Drug: Crisaborole ointment, 2% — Applied twice a day (BID)
  Other Names: Eucrisa
  Arms: Crisaborole ointment, 2%
Drug: Hydrocortisone butyrate cream, 0.1% — Applied BID
  Other Names: Locoid 0.1%
  Arms: Hydrocortisone butyrate cream, 0.1%
Drug: Pimecrolimus cream, 1% — Applied BID
  Other Names: Elidel
  Arms: Pimecrolimus cream, 1%
Drug: Crisaborole Vehicle — Applied BID
  Arms: Crisaborole Vehicle

SUMMARY:
This 4-week study will evaluate the safety and efficacy of crisaborole ointment 2%; crisaborole vehicle; topical corticosteroid and topical calcineurin inhibitor, applied twice daily (BID) in subjects who are at least 2 years of age with mild-moderate AD.

A Sub-Study of Optical Coherence Tomography and Biomarkers in Subjects ages 2 to <18 years old, with Mild to Moderate Atopic Dermatitis, treated with Crisaborole Ointment, 2% or Crisaborole Vehicle Ointment or Hydrocortisone Butyrate 0.1% Cream applied BID will also be conducted at select sites.

DETAILED DESCRIPTION:
Approximately 600 subjects will be enrolled in the study, of which at least 150 subjects aged 2-6; at least 140 subjects aged 7-11; at least 120 subjects aged 12-17 and up to 90 subjects will be adults. Subjects must have mild-moderate AD involving at least 5% treatable %BSA assessed on baseline/Day 1. Treatable %BSA will be defined as the percent of a subject's total body surface area that is AD involved, excluding the scalp.

Eligible subjects will be randomized at the Baseline/Day 1 visit. Randomization will be stratified by eligibility for TCS or TCI treatment as per national approved labels. Cohort 1 will be for subjects who are eligible for TCS therapy, and Cohort 2 will be for subjects who are not eligible for TCS therapy but eligible for TCI therapy. The investigational products will be applied BID for 28 days to the Treatable body surface area (BSA) identified at Baseline/Day 1.

The primary efficacy endpoint is the percent change from baseline in the Eczema Area and Severity Index (EASI) total score at Day 29.

For the efficacy comparison of crisaborole versus vehicle, subjects from both Cohort 1 and Cohort 2 are included in the analysis, adjusted for cohort effect. For the efficacy comparison of crisaborole versus TCS, only subjects from Cohort 1 are included in the analysis. For the comparison of crisaborole versus TCI, only subjects from Cohort 2 are included in the analysis.

Safety and efficacy assessments will be conducted at the investigator site by a clinical assessor blinded to treatment assignment.

Scheduled study visits for all subjects will occur at Screening, Baseline/Day 1, Day 8, Day 15, Day 22, Day 29 (End of treatment/Early termination), Day 43 or 14 Days after last dose if subject is terminated early from treatment. A follow up telephone call will be made by site staff to the subjects/subject's legally acceptable guardian(s) on Day 60 or at least 28 days after last dose if subject is terminated early from treatment. The Day 60 visit will be completed in the clinic for subjects enrolled in the OCT sub-study.

To further explore the benefit/risk of crisaborole ointment, 2%, a sub-study to evaluate differences in atrophic skin changes across study treatment groups in Cohort 1 will be conducted at select sites.

The sub-study will include obtaining Optical coherence tomography (OCT) imaging to evaluate atrophic changes in epidermal thickness during and after treatment with study investigational product in Cohort 1. This sub-study also provides an opportunity to explore differences in Transepidermal Water Loss (TEWL) and cutaneous inflammatory and barrier biomarkers associated with AD within the stratum corneum (SC) across treatment groups in Cohort 1. The Aquaflux (an evaporimeter) will be used in this sub-study to evaluate TEWL during and after treatment at select sub-study centers. Tape-strips will also be used in this sub-study to evaluate SC biomarkers from AD lesional and non-lesional skin.

This sub-study will include approximately 60 subjects from Cohort 1 that are enrolled in the main study (C3291037). Subjects will follow the main study assessments and visits as per the schedule of activities for the main study but will also follow additional procedures as described in the protocol. The telephone call at Day 60 in the main study is replaced with an in-clinic visit for sub-study participants.

ELIGIBILITY:
Inclusion Criteria:

Is male or female 2 years and older at the Screening visit/time of informed consent/assent diagnosed with mild-moderate AD (according to the criteria of Hanifin and Rajka), of at least 5% BSA.

Exclusion Criteria:

Has any clinically significant medical disorder, condition, or disease (including active or potentially recurrent non AD dermatological conditions and known genetic dermatological conditions that overlap with AD, such as Netherton syndrome.

Subjects in Cohort 1 are excluded if they have a contraindication for treatment with hydrocortisone butyrate cream 0.1%

Subjects in Cohort 2 are excluded if they have a contraindication for treatment with pimecrolimus cream, 1%

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (32):
- United States (10):
  - Dermatology Trial Associates, Bryant, Arkansas
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Park Avenue Dermatology, Orange Park, Florida
  - Lenus Research & Medical Group, LLC, Sweetwater, Florida
  - ForCare Clinical Research, Tampa, Florida
  - DS Research, Louisville, Kentucky
  - M3-Wake Research, Inc., Raleigh, North Carolina
  - Arlington Research Center, Inc., Arlington, Texas
  - Tanner Clinic, Layton, Utah
  - Virginia Clinical Research, Inc, Norfolk, Virginia
- Germany (6):
  - Klinikum der Universitat Munchen, München, Bavaria
  - Fachklinik Bad Bentheim, Fachbereich Dermatologie und Allergologie, Dermatologische Ambulanz, Bad Bentheim, Lower Saxony
  - Universitatsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitatsklinikum Schleswig-Holstein, Campus Lubeck, Lübeck, Schleswig-Holstein
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - Universitaetsklinikum Frankfurt, Frankfurt am Main
- Italy (4):
  - UOSD Dermatologia Gen. ed Oncologica DU, PO San Salvatore, L’Aquila, AQ
  - DiSSal Sezione di Dermatologia Az. Ospedaliera Universitaria, Genova, GE
  - Ospedale San Pietro Fatebenefratelli, Roma, RM
  - Azienda Ospedaliero - Universitaria Policlinico Tor Vergata, Roma, ROME
- Poland (5):
  - Barbara Rewerska Diamond Clinic, Krakow, Malopolska
  - Silmedic sp. z o.o, Katowice
  - Krakowskie Centrum Medyczne sp. z o.o., Krakow
  - Klinika Ambroziak Sp. z O. O., Warsaw
  - ROYALDERM Agnieszka Nawrocka, Warsaw
- Sweden (2):
  - Barn och Ungdomskliniken, Örebro
  - Avdelningen for Kliniska Provningar, Örebro
- Switzerland (3):
  - Universitatsklinik fuer Dermatologie, Bern
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - Universitats-Kinderspital Zurich, Zurich
- United Kingdom (2):
  - Rame Medical Ltd, Penntorr Health, Torpoint, Cornwall
  - NHS Tayside, Ninewells Hospital and Medical School, Dundee, Scotland

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3291037

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At time of early termination, less than 40% of planned participants were treated across treatment groups. Number of participants enrolled up to early termination of study were insufficient to allow a meaningful inference and robust statistical analyses of data. As a result, all safety data was summarized with Cohort 1 and Cohort 2 combined for crisaborole and vehicle groups.
Pre-assignment Details: This study was originally plan to conduct in 2 different cohorts for crisaborole and vehicle groups. Cohort 1 was planned for participants eligible for topical corticosteroid (TCS) therapy (hydrocortisone butyrate cream 0.1%), and Cohort 2 was planned for participants not eligible for TCS therapy but eligible for topical calcineurin inhibitor (TCI) therapy (pimecrolimus cream 1%).
Groups:
- Vehicle: Vehicle matched to crisaborole 2% ointment was applied topically bis in diem (BID - twice a day) to all treatable atopic dermatitis (AD) involved areas (excluding the scalp) identified at Baseline (Day 1) through Day 28. End of treatment visit was scheduled on Day 29. Participants were followed-up for at least 28 days after last dose, maximum up to Day 60.
- Crisaborole Ointment 2% BID: Crisaborole ointment 2% was applied topically BID to all treatable AD involved areas (excluding the scalp) identified at Baseline (Day 1) through Day 28. End of treatment visit was scheduled on Day 29. Participants were followed-up for at least 28 days after last dose, maximum up to Day 60.
- Hydrocortisone Butyrate Cream 0.1% BID: Hydrocortisone butyrate cream 0.1% was applied topically BID to all treatable AD involved areas (excluding the scalp) identified at Baseline (Day 1) through Day 28. End of treatment visit was scheduled on Day 29. Participants were followed-up for at least 28 days after last dose, maximum up to Day 60.
- Pimecrolimus Cream 1% BID: Pimecrolimus cream 1% was applied topically BID to all treatable AD involved areas (excluding the scalp) identified at Baseline (Day 1) through Day 28. End of treatment visit was scheduled on Day 29. Participants were followed-up for at least 28 days after last dose, maximum up to Day 60.
Period: Overall Study
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Started | 60 | 59 | 71 | 47
Treated | 59 | 58 | 71 | 47
Completed | 54 | 52 | 65 | 46
Not Completed | 6 | 7 | 6 | 1
Not completed — Withdraw by parent/guardian | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 2 | 4 | 5 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1
Not completed — Randomized but not treated | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants received at least 1 dose of investigational product.
Groups:
- Vehicle: Vehicle matched to crisaborole 2% ointment was applied topically BID to all treatable AD involved areas (excluding the scalp) identified at Baseline (Day 1) through Day 28. End of treatment visit was scheduled on Day 29. Participants were followed-up for at least 28 days after last dose, maximum up to Day 60.
- Total: Total of all reporting groups
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID | Total
Number analyzed (Participants) | 59 | 58 | 71 | 47 | 235
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19.8 (18.22) | 21.5 (19.12) | 19.6 (16.28) | 21.1 (18.20) | 20.4 (17.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 43 | 26 | 139
  Male | 24 | 23 | 28 | 21 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 11 | 4 | 22
  Not Hispanic or Latino | 53 | 57 | 60 | 43 | 213
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 1 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 17 | 14 | 23 | 6 | 60
  White | 38 | 38 | 44 | 37 | 157
  More than one race | 1 | 3 | 1 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in the Eczema Area and Severity Index (EASI) Total Score at Day 29
Description: EASI quantifies severity of participant's AD (excluded scalp) based on lesion severity and percent (%) body surface area (%BSA) affected. Lesion severity included erythema (E), induration/papulation (I), excoriation (Ex), lichenification (L) scored for 4 regions (head and neck [h], upper limbs [u], trunk [t] [including axillae, groin], lower limbs [l] [including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score (A) based upon %BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%), 6 (90 to 100%). Total EASI score (aged >=8 years) =0.1*Ah*(Eh + Ih + Exh + Lh) + 0.2*Au*(Eu + Iu + Exu + Lu) + 0.3*At*(Et + It +Ext + Lt) + 0.4*Al*(El + Il + Exl + Ll); for aged 2 to <8 years =0.2*Ah*(Eh + Ih + Exh + Lh) + 0.2*Au*(Eu + Iu + Exu + Lu) + 0.3*At*(Et +It + Ext + Lt) + 0.3*Al*(El + Il + Exl + Ll). Total score ranges from 0.0 to 72.0, higher scores indicated greater AD severity.
Time Frame: Baseline, Day 29
Population: FAS included all randomized participants who received at least 1 dose of investigational product. Here, "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Vehicle: Participants 2-17 Years; Vehicle: Participants >=18 Years: Vehicle matched to crisaborole 2% ointment was applied topically BID to all treatable AD involved areas (excluding the scalp) identified at Baseline (Day 1) through Day 28. End of treatment visit was scheduled on Day 29. Participants were followed-up for at least 28 days after last dose, maximum up to Day 60.
- Crisaborole Ointment 2% BID: Participants 2-17 Years; Crisaborole Ointment 2% BID: Participants >=18 Years: Crisaborole ointment 2% was applied topically BID to all treatable AD involved areas (excluding the scalp) identified at Baseline (Day 1) through Day 28. End of treatment visit was scheduled on Day 29. Participants were followed-up for at least 28 days after last dose, maximum up to Day 60.
- Hydrocortisone Butyrate Cream 0.1% BID: Participants 2-17 Years; Hydrocortisone Butyrate Cream 0.1% BID: Participants >=18 Years: Hydrocortisone butyrate cream 0.1% was applied topically BID to all treatable AD involved areas (excluding the scalp) identified at Baseline (Day 1) through Day 28. End of treatment visit was scheduled on Day 29. Participants were followed-up for at least 28 days after last dose, maximum up to Day 60.
- Pimecrolimus Cream 1% BID: Participants 2-17 Years; Pimecrolimus Cream 1% BID: Participants >=18 Years: Pimecrolimus cream 1% was applied topically BID to all treatable AD involved areas (excluding the scalp) identified at Baseline (Day 1) through Day 28. End of treatment visit was scheduled on Day 29. Participants were followed-up for at least 28 days after last dose, maximum up to Day 60.
Arm/Group | Vehicle: Participants 2-17 Years | Crisaborole Ointment 2% BID: Participants 2-17 Years | Hydrocortisone Butyrate Cream 0.1% BID: Participants 2-17 Years | Pimecrolimus Cream 1% BID: Participants 2-17 Years | Vehicle: Participants >=18 Years | Crisaborole Ointment 2% BID: Participants >=18 Years | Hydrocortisone Butyrate Cream 0.1% BID: Participants >=18 Years | Pimecrolimus Cream 1% BID: Participants >=18 Years
Number analyzed (Participants) | 31 | 31 | 36 | 29 | 17 | 19 | 29 | 14
Percent change | -26.62 (46.283) | -49.47 (34.195) | -75.50 (30.305) | -60.08 (31.877) | -44.67 (49.267) | -57.14 (48.345) | -70.29 (32.097) | -62.59 (28.317)

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Treatment Discontinuations Due to AEs and SAEs
Description: An AE is any untoward medical occurrence in a study participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. TEAEs are events between the first dose of study drug up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. A SAE is any untoward medical occurrence at any dose that: results in death; is life-threatening (immediate risk of death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); results in congenital anomaly/birth defect; or that is considered to be an important medical event.
Time Frame: From Baseline up to 28 days after last dose of study treatment (maximum up to 60 Days)
Population: Safety analysis set included all participants who received at least 1 dose of the investigational product according to actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 59 | 58 | 71 | 47
Participants
  TEAEs | 18 | 25 | 12 | 24
  SAEs | 0 | 0 | 0 | 0
  Discontinuation due to AEs | 0 | 3 | 0 | 0
  Discontinuation due to SAEs | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Local Tolerability Adverse Events (AEs)
Description: Local tolerability AEs included application and instillation site reactions, application site discharge, application site erythema, application site exfoliation, application site pain, application site pruritus, application site swelling, dermatitis and eczema, dermatitis atopic, dermatitis contact, eczema, skin irritation, telangiectasia and related conditions, and urticarias.
Time Frame: From Baseline up to 28 days after last dose of study treatment (maximum up to 60 Days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 59 | 58 | 71 | 47
Participants | 12 | 13 | 2 | 8

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Vital sign measurements included temperature, respiratory rate, pulse rate, and blood pressure. Temperature, respiratory rate, pulse rate, and blood pressure were taken in the seated or supine position, after the participant has been sitting or lying calmly for a minimum of 5 minutes (when possible for younger children). Position of recording was consistent within participant through-out the study.
Time Frame: Screening up to Day 29
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 59 | 58 | 71 | 47
Participants | 0 | 0 | 1 | 0

5. Secondary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Total Score at Day 8, 15 and 22
Description: EASI quantifies severity of participant's AD (excluded scalp) based on lesion severity and %BSA affected. Lesion severity included erythema (E), induration/papulation (I), excoriation (Ex), lichenification (L) scored for 4 regions (head and neck [h], upper limbs [u], trunk [t] [including axillae, groin], lower limbs [l] [including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score(A) based upon %BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%), 6 (90 to 100%). Total EASI score (aged >=8 years) =0.1*Ah*(Eh + Ih + Exh + Lh) + 0.2*Au*(Eu + Iu + Exu + Lu) + 0.3*At*(Et + It +Ext + Lt) + 0.4*Al*(El + Il + Exl + Ll); for aged 2 to <8 years =0.2*Ah*(Eh + Ih + Exh + Lh) + 0.2*Au*(Eu + Iu + Exu + Lu) + 0.3*At*(Et +It + Ext + Lt) + 0.3*Al*(El + Il + Exl + Ll). Total score ranges from 0.0 to 72.0, higher scores indicated greater AD severity.
Time Frame: Baseline, Day 8, 15 and 22
Population: FAS included all randomized participants who received at least 1 dose of investigational product. Here, 'number analyzed' signifies number of participants evaluable for each specified row.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Vehicle: Participants 2-17 Years | Crisaborole Ointment 2% BID: Participants 2-17 Years | Hydrocortisone Butyrate Cream 0.1% BID: Participants 2-17 Years | Pimecrolimus Cream 1% BID: Participants 2-17 Years | Vehicle: Participants >=18 Years | Crisaborole Ointment 2% BID: Participants >=18 Years | Hydrocortisone Butyrate Cream 0.1% BID: Participants >=18 Years | Pimecrolimus Cream 1% BID: Participants >=18 Years
Number analyzed (Participants) | 38 | 37 | 38 | 30 | 21 | 21 | 32 | 17
Percent change
  Percent Change at Day 8: number analyzed (Participants) | 37 | 33 | 33 | 29 | 19 | 21 | 27 | 16
  Percent Change at Day 8 | -17.88 (36.705) | -26.79 (39.280) | -45.59 (28.103) | -34.20 (25.972) | -14.77 (26.308) | -29.83 (44.599) | -42.48 (27.843) | -18.75 (39.016)
  Percent Change at Day 15: number analyzed (Participants) | 33 | 33 | 37 | 30 | 15 | 20 | 27 | 14
  Percent Change at Day 15 | -25.77 (35.658) | -36.72 (36.625) | -58.96 (32.617) | -42.75 (31.854) | -25.93 (31.690) | -48.42 (33.458) | -56.29 (32.186) | -37.18 (50.487)
  Percent Change at Day 22: number analyzed (Participants) | 32 | 31 | 35 | 26 | 18 | 19 | 27 | 15
  Percent Change at Day 22 | -25.07 (49.326) | -38.87 (32.624) | -69.09 (31.528) | -59.86 (24.835) | -34.43 (30.587) | -56.05 (38.934) | -61.82 (27.894) | -42.25 (40.192)

6. Secondary Outcome: Number of Participants Who Achieved Success in the Investigator's Static Global Assessment (ISGA) (ISGA Score of Clear [0] or Almost Clear [1] With At-least a 2-Grade Improvement From Baseline) at Day 8, 15, 22 and 29
Description: ISGA is a five point global assessment scale of AD severity, used to characterize participants' overall disease severity across all treatable AD lesions (excluding the scalp). ISGA score ranged from 0 to 4: where 0= clear (minor residual hypo/hyperpigmentation; no erythema or induration/papulation; no oozing/crusting), 1= almost clear (trace faint pink erythema, with barely perceptible induration/papulation and no oozing/crusting), 2= mild (faint pink erythema with mild induration/papulation and no oozing/crusting), 3= moderate (pink-red erythema with moderate induration/papulation with or without oozing/crusting), 4= severe (deep or bright red erythema with severe induration/papulation and with oozing/crusting). Higher scores indicated greater severity of AD.
Time Frame: Day 8, 15, 22 and 29
Population: FAS included all randomized participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle: Participants 2-17 Years | Crisaborole Ointment 2% BID: Participants 2-17 Years | Hydrocortisone Butyrate Cream 0.1% BID: Participants 2-17 Years | Pimecrolimus Cream 1% BID: Participants 2-17 Years | Vehicle: Participants >=18 Years | Crisaborole Ointment 2% BID: Participants >=18 Years | Hydrocortisone Butyrate Cream 0.1% BID: Participants >=18 Years | Pimecrolimus Cream 1% BID: Participants >=18 Years
Number analyzed (Participants) | 38 | 37 | 39 | 30 | 21 | 21 | 32 | 17
Participants
  Day 8 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Day 15 | 1 | 3 | 8 | 2 | 0 | 0 | 6 | 1
  Day 22 | 2 | 2 | 11 | 5 | 1 | 3 | 9 | 1
  Day 29 | 2 | 5 | 20 | 7 | 3 | 6 | 13 | 2

7. Secondary Outcome: Number of Participants Who Achieved Investigator's Static Global Assessment (ISGA) Score of Clear (0) or Almost Clear (1) at Day 8, 15, 22 and 29
Description: ISGA is a five point global assessment scale of AD severity, used to characterize participants' overall disease severity across all treatable AD lesions (excluding the scalp). ISGA score ranged from 0 to 4: where 0 = clear (minor residual hypo/hyperpigmentation; no erythema or induration/papulation; no oozing/crusting), 1= almost clear (trace faint pink erythema, with barely perceptible induration/papulation and no oozing/crusting), 2= mild (faint pink erythema with mild induration/papulation and no oozing/crusting), 3= moderate (pink-red erythema with moderate induration/papulation with or without oozing/crusting), 4= severe (deep or bright red erythema with severe induration/papulation and with oozing/crusting). Higher scores indicated greater severity of AD.
Time Frame: Day 8, 15, 22 and 29
Population: FAS included all randomized participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle: Participants 2-17 Years | Crisaborole Ointment 2% BID: Participants 2-17 Years | Hydrocortisone Butyrate Cream 0.1% BID: Participants 2-17 Years | Pimecrolimus Cream 1% BID: Participants 2-17 Years | Vehicle: Participants >=18 Years | Crisaborole Ointment 2% BID: Participants >=18 Years | Hydrocortisone Butyrate Cream 0.1% BID: Participants >=18 Years | Pimecrolimus Cream 1% BID: Participants >=18 Years
Number analyzed (Participants) | 38 | 37 | 39 | 30 | 21 | 21 | 32 | 17
Participants
  Day 8 | 6 | 3 | 12 | 5 | 0 | 4 | 4 | 2
  Day 15 | 6 | 7 | 19 | 9 | 1 | 3 | 11 | 5
  Day 22 | 6 | 8 | 19 | 9 | 1 | 8 | 13 | 5
  Day 29 | 6 | 10 | 27 | 13 | 4 | 9 | 20 | 7

8. Secondary Outcome: Number of Participants Who Achieved Greater Than or Equal to (>=) 75 Percent (%) Improvement From Baseline in Eczema Area and Severity Index (EASI) Total Score at Day 8, 15, 22 and 29
Description: as for outcome 5
Time Frame: Day 8, 15, 22 and 29
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 59 | 58 | 70 | 47
Participants
  Day 8 | 2 | 7 | 9 | 2
  Day 15 | 4 | 10 | 25 | 8
  Day 22 | 8 | 13 | 29 | 11
  Day 29 | 9 | 17 | 40 | 17

9. Secondary Outcome: Time to First Improvement From Baseline in Eczema Area and Severity Index (EASI) Total Score of Greater Than or Equal to (>=) 75%
Description: as for outcome 5
Time Frame: Baseline up to Day 43
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 59 | 58 | 70 | 47
Days | NA [NA to NA] — Median and 95% CI could not be estimated because there were insufficient number of participants with event. | 43.0 [28.0 to NA] — Upper limit for 95% CI could not be estimated because there were insufficient number of participants with events to calculate the full 95% CI. | 23.0 [16.0 to 34.0] | 32.0 [27.0 to NA] — Upper limit for 95% CI could not be estimated because there were insufficient number of participants with events to calculate the full 95% CI.

10. Secondary Outcome: Change From Baseline in Percent Body Surface Area (%BSA) at Day 8, 15, 22 and 29
Description: Four body regions were evaluated: head and neck, upper limbs, trunk (including axillae) and lower limbs (including buttocks) excluding scalp. BSA was calculated using handprint method. Number of handprints (size of participant's full palmer hand in a closed position) fitting in affected area of a body region was estimated. Maximum number of handprints were: 10 for head, neck (20 for <8 years age), 20 for upper limbs, 30 for trunk, 40 for lower limbs (30 for <8 years age). Surface area (SA) of body region equivalent to 1 handprint: 10% for head, neck (5% for <8 years age), 5% for upper limbs, 3.33% for trunk, 2.5% for lower limbs (3.33% for <8 years age). Overall %BSA for a body region = total number of handprints in a body region * % SA equivalent to 1 handprint. % BSA for an individual: mean of % BSA of all 4 body regions, range =0-100%, higher values = greater AD severity.
Time Frame: Baseline, Day 8, 15, 22 and 29
Population: FAS included all randomized participants who received at least 1 dose of investigational product. Here 'number analyzed' signifies number of participants evaluable for each specified row.
Measure: Mean (Standard Deviation); unit: Percent BSA
Arm/Group | Vehicle: Participants 2-17 Years | Crisaborole Ointment 2% BID: Participants 2-17 Years | Hydrocortisone Butyrate Cream 0.1% BID: Participants 2-17 Years | Pimecrolimus Cream 1% BID: Participants 2-17 Years | Vehicle: Participants >=18 Years | Crisaborole Ointment 2% BID: Participants >=18 Years | Hydrocortisone Butyrate Cream 0.1% BID: Participants >=18 Years | Pimecrolimus Cream 1% BID: Participants >=18 Years
Number analyzed (Participants) | 38 | 37 | 39 | 30 | 21 | 21 | 32 | 17
Percent BSA
  Change at Day 8: number analyzed (Participants) | 37 | 33 | 33 | 29 | 19 | 21 | 27 | 16
  Change at Day 8 | -2.04 (7.533) | -2.63 (11.920) | -5.25 (8.346) | -2.84 (5.296) | -1.39 (4.417) | -4.09 (6.397) | -2.74 (2.718) | -1.44 (5.600)
  Change at Day 15: number analyzed (Participants) | 33 | 33 | 37 | 30 | 15 | 20 | 27 | 14
  Change at Day 15 | -2.38 (8.566) | -4.32 (12.620) | -7.40 (9.515) | -3.72 (4.401) | -3.73 (5.895) | -4.63 (7.211) | -5.00 (5.189) | -3.56 (5.750)
  Change at Day 22: number analyzed (Participants) | 32 | 31 | 35 | 26 | 18 | 19 | 27 | 15
  Change at Day 22 | -2.23 (12.321) | -7.14 (10.123) | -8.54 (11.226) | -6.52 (9.883) | -4.19 (5.464) | -5.98 (7.852) | -4.91 (5.190) | -4.17 (5.588)
  Change at Day 29: number analyzed (Participants) | 31 | 31 | 36 | 29 | 17 | 19 | 29 | 14
  Change at Day 29 | -3.38 (9.974) | -9.95 (11.324) | -9.63 (12.309) | -7.30 (10.774) | -6.76 (8.089) | -7.18 (8.183) | -7.18 (5.971) | -6.86 (8.172)

11. Secondary Outcome: Change From Baseline in Peak Pruritus Numerical Rating Scale (NRS) in Participants Aged Greater Than or Equal to (>=) 12 Years at Day 8, 15, 22 and 29
Description: The severity of itch (pruritus) due to AD was assessed using the peak pruritus NRS for participants aged >=12 years. Participants at specified time points were asked the following question: "how would you rate your itch at the worst moment during the previous 24 hours?" The scale ranged from 0 to 10, where 0= no itch and 10= worst itch imaginable. Higher scores indicated worse itch.
Time Frame: Baseline, Day 8, 15, 22 and 29
Population: Analysis was performed on all participants aged >=12 years from FAS, and FAS included all randomized participants who received at least 1 dose of investigational product. Here, "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure and 'number analyzed' signifies number of participants evaluable for each specified row.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 33 | 33 | 45 | 28
Units on a scale
  Change at Day 8: number analyzed (Participants) | 30 | 30 | 43 | 26
  Change at Day 8 | -0.67 (1.254) | -1.01 (1.145) | -2.24 (2.065) | -0.29 (1.225)
  Change at Day 15: number analyzed (Participants) | 29 | 32 | 43 | 25
  Change at Day 15 | -0.97 (1.778) | -1.08 (1.419) | -3.21 (2.598) | -1.35 (1.707)
  Change at Day 22: number analyzed (Participants) | 27 | 30 | 42 | 24
  Change at Day 22 | -0.98 (1.887) | -1.28 (1.642) | -3.83 (2.554) | -1.66 (1.759)
  Change at Day 29: number analyzed (Participants) | 27 | 29 | 42 | 24
  Change at Day 29 | -1.30 (2.157) | -1.65 (1.996) | -4.02 (2.734) | -1.67 (1.952)

12. Secondary Outcome: Change From Baseline in Participant Reported Itch Severity Scale in Participants Aged 6-11 Years at Day 8, 15, 22 and 29
Description: The severity of itch (pruritus) due to AD was assessed using the five-category participant reported itch severity scale for participants aged 6-11 years. Participants at specified time points were asked to "circle the face that shows how itchy your skin has been today". The scale ranged from 0 to 4, where 0= no itch and 4= very itch. Higher scores indicated worse itch.
Time Frame: Baseline, Day 8, 15, 22 and 29
Population: Data was not summarized as per SAP which was revised prior to the analyses and which reflect limitations related to reduced sample size (39% enrollment) of early terminated study. Smaller than originally planned sample size was insufficient to allow robust statistical analyses. Pruritus related PRO endpoints used different instruments in each of 3 age groups. As a result, subdividing population based on age group renders smaller sample size in pediatric groups, therefore data was not summarized.
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Change From Baseline in Observer Reported Itch Severity Scale in Participants Aged Less Than (<) 6 Years at Day 8, 15, 22 and 29
Description: The severity of itch (pruritus) due to AD was assessed using the participant reported itch severity scale for participants aged <6 years. Participant's caregivers at specified time points were asked the following question "how would you rate your observation of your child's itch (scratching, rubbing) at the worst moment during the previous 24 hours?". The scale ranged from 0 to 10, where 0= no itch and 10= worst itch imaginable. Higher scores indicated worse itch.
Time Frame: Baseline, Day 8, 15, 22 and 29
Population: as for outcome 12
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Time to Greater Than or Equal to (>=2) Point Improvement From Baseline in Peak Pruritus Numeric Rating Scale (NRS) in Participants Aged Greater Than (>) 12 Years
Description: The severity of itch (pruritus) due to AD was assessed using the peak pruritus NRS for participants aged >12 years. Participants at specified time points were asked the following question: "how would you rate your itch at the worst moment during the previous 24 hours?" The scale ranged from 0 to 10, where 0= no itch and 10= worst itch imaginable. Higher scores indicated worse itch.
Time Frame: Baseline up to Day 29
Population: Data was not summarized as per SAP which was revised prior to the analyses and which reflected limitations related to reduced sample size (only 39% enrollment) of early terminated study. Smaller than originally planned sample size was insufficient to allow robust statistical analyses. Summarizing further by Time to >2 Point Improvement will not provide additional useful information due to smaller than planned sample size as a result of study early termination.
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Time to >= 3 Point Improvement From Baseline in Peak Pruritus Numeric Rating Scale (NRS) in Participants Aged Greater Than (>)12 Years
Description: as for outcome 14
Time Frame: Baseline up to Day 29
Population: Data was not summarized as per SAP which was revised prior to the analyses and which reflected limitations related to reduced sample size (only 39% enrollment) of early terminated study. Smaller than originally planned sample size was insufficient to allow robust statistical analyses. Summarizing further by Time to >3 Point Improvement will not provide additional useful information due to smaller than planned sample size as a result of study early termination.
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Secondary Outcome: Time >=2 Point to Improvement From Baseline in Observer Reported Itch Severity Scale in Participants Aged Less Than (<) 6 Years
Description: The severity of itch (pruritus) due to AD was assessed using the patient reported itch severity scale for participants aged <6 years. Participant's caregivers at specified time points were asked the following question "how would you rate your observation of your child's itch (scratching, rubbing) at the worst moment during the previous 24 hours?". The scale ranged from 0 to 10, where 0= no itch and 10= worst itch imaginable. Higher scores indicated worse itch.
Time Frame: Baseline up to Day 29
Population: as for outcome 12
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Time to >=3 Point Improvement From Baseline in Observer Reported Itch Severity Scale in Participants Aged Less Than (<) 6 Years
Description: as for outcome 16
Time Frame: Baseline up to Day 29
Population: as for outcome 12
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants Who Achieved >=2 Point Improvement From Baseline in Peak Pruritus Numeric Rating Scale (NRS) in Participants Aged Greater Than or Equal to (>=) 12 Years at Day 8, 15, 22 and 29
Description: as for outcome 11
Time Frame: Day 8, 15, 22 and 29
Population: Analysis was performed on all participants aged >=12 years from FAS, and FAS included all randomized participants who received at least 1 dose of investigational product. Here, "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 31 | 32 | 42 | 26
Participants
  Day 8 | 3 | 7 | 21 | 1
  Day 15 | 9 | 8 | 31 | 7
  Day 22 | 9 | 7 | 32 | 9
  Day 29 | 10 | 9 | 32 | 9

19. Secondary Outcome: Number of Participants Who Achieved >=3 Point Improvement From Baseline in Peak Pruritus Numeric Rating Scale (NRS) in Participants Aged Greater Than or Equal to (>=) 12 Years at Day 8, 15, 22 and 29
Description: as for outcome 11
Time Frame: Day 8, 15, 22 and 29
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 29 | 29 | 40 | 26
Participants
  Day 8 | 2 | 1 | 11 | 0
  Day 15 | 5 | 5 | 21 | 3
  Day 22 | 4 | 4 | 25 | 4
  Day 29 | 6 | 6 | 24 | 6

20. Secondary Outcome: Number of Participants Who Achieved Greater Than or Equal to (>=) 2 Point Improvement From Baseline in Observer Reported Itch Severity Scale in Participants Aged Less Than (<) 6 Years at Day 8, 15, 22 and 29
Description: as for outcome 16
Time Frame: Day 8, 15, 22 and 29
Population: as for outcome 12
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Participants Who Achieved Greater Than or Equal to (>=) 3 Point Improvement From Baseline in Observer Reported Itch Severity Scale in Participants Aged Less Than (<) 6 Years at Day 8, 15, 22 and 29
Description: as for outcome 16
Time Frame: Day 8, 15, 22 and 29
Population: as for outcome 12
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 0 | 0 | 0 | 0

22. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) in Participants Greater Than or Equal to (>=) 16 Years at Day 8, 15, 22 and 29
Description: DLQI is a 10-item questionnaire that measures the impact of skin disease on participants aged >=16 years. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicated more impact on quality of life. Scores from all 10 questions were added up to give DLQI total score range from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of participant.
Time Frame: Baseline, Day 8, 15, 22 and 29
Population: Analysis was performed on all participants aged >=16 years from FAS, and FAS included all randomized participants who received at least 1 dose of investigational product. Here, "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure and 'number analyzed' signifies number of participants evaluable for each specified row.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 23 | 26 | 32 | 23
Units on a scale
  Change at Day 8: number analyzed (Participants) | 20 | 23 | 27 | 19
  Change at Day 8 | -1.9 (5.53) | -3.8 (3.45) | -5.1 (4.98) | -1.4 (2.99)
  Change at Day 15: number analyzed (Participants) | 16 | 23 | 26 | 17
  Change at Day 15 | -3.4 (3.72) | -3.5 (2.92) | -6.8 (5.94) | -2.9 (2.63)
  Change at Day 22: number analyzed (Participants) | 18 | 20 | 25 | 18
  Change at Day 22 | -2.8 (4.12) | -3.4 (4.73) | -6.9 (6.37) | -3.4 (3.88)
  Change at Day 29: number analyzed (Participants) | 18 | 19 | 28 | 17
  Change at Day 29 | -4.9 (5.60) | -3.9 (4.76) | -7.0 (6.69) | -4.1 (3.76)

23. Secondary Outcome: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) in Participants Aged 4-15 Years at Day 8, 15, 22 and 29
Description: The CDLQI was a 10-item questionnaire that measures the impact of skin disease on children's (aged 4 to 15 years) quality of life. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. The CDLQI total score was the sum of individual scores of question 1-10 and ranged from 0 (not at all) to 30 (very much): 0-1 = no effect on the child's life; 2-6 = small effect; 7-12 = moderate effect; 13-18 = very large effect; 19-30 = extremely large effect. Higher scores indicated more impact on quality of life of children.
Time Frame: Baseline, Day 8, 15, 22 and 29
Population: Analysis was performed on all participants aged 4 to 15 years from FAS, and FAS included all randomized participants who received at least 1 dose of investigational product. Here, "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure and 'number analyzed' = participants evaluable for each specified row.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 27 | 26 | 30 | 18
Units on a scale
  Change at Day 8: number analyzed (Participants) | 27 | 22 | 25 | 15
  Change at Day 8 | -0.2 (3.42) | -2.1 (4.49) | -5.4 (6.14) | -1.7 (4.03)
  Change at Day 15: number analyzed (Participants) | 22 | 24 | 29 | 17
  Change at Day 15 | -2.0 (4.49) | -3.1 (5.13) | -5.5 (6.32) | -1.6 (4.66)
  Change at Day 22: number analyzed (Participants) | 21 | 21 | 27 | 13
  Change at Day 22 | -2.7 (3.04) | -2.6 (5.81) | -4.9 (7.89) | -2.5 (3.15)
  Change at Day 29: number analyzed (Participants) | 20 | 21 | 28 | 16
  Change at Day 29 | -3.1 (2.73) | -3.4 (4.85) | -6.4 (5.49) | -3.4 (3.52)

24. Secondary Outcome: Change From Baseline in Dermatitis Family Impact Questionnaire (DFI) in Participants Aged 2-17 Years at Day 8, 15, 22 and 29
Description: The DFI was a 10-item disease questionnaire that measures the impact of having a child (aged 2-17 years) with AD on family quality of life. It was completed by parent/legal guardian of the child (affected by AD), based on recall over the past week. Each question was scored on a 4-point scale ranging from 0 (not at all) to 30 (very much): where higher scores indicated worst quality of life of family. The DFI total score was the sum of individual scores of the 10 questions and ranged from 0 (no impact on life of family) to 30 (maximum effect on life of family), where higher DFI scores indicated maximum effect on life of family.
Time Frame: Baseline, Day 8, 15, 22 and 29
Population: Analysis was performed on all participants aged 2 to 17 years from FAS, and FAS included all randomized participants who received at least 1 dose of investigational product. Here, "Overall Number of Participants Analyzed" = participants evaluable for this outcome measure and 'number analyzed' = participants evaluable for each specified row.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 38 | 37 | 39 | 30
Units on a scale
  Change at Day 8: number analyzed (Participants) | 37 | 32 | 33 | 28
  Change at Day 8 | -1.2 (6.43) | -2.3 (5.16) | -5.6 (5.61) | -2.8 (6.79)
  Change at Day 15: number analyzed (Participants) | 32 | 31 | 37 | 30
  Change at Day 15 | -1.1 (6.77) | -2.3 (4.71) | -5.5 (6.82) | -3.2 (5.94)
  Change at Day 22: number analyzed (Participants) | 31 | 29 | 34 | 26
  Change at Day 22 | -2.5 (4.84) | -3.1 (5.24) | -5.3 (6.92) | -4.5 (5.93)
  Change at Day 29: number analyzed (Participants) | 30 | 28 | 35 | 29
  Change at Day 29 | -1.8 (5.26) | -3.6 (4.40) | -6.4 (5.61) | -4.8 (5.61)

25. Primary Outcome: Number of Participants With Clinically Significant Abnormal Laboratory Parameters
Description: Hematology parameters included with criteria greater than (>) 1.2*upper limit of normal (ULN): leukocytes (10^3 per cubic millimeter [10^3/mm^3]), lymphocytes (10^3/mm^3), lymphocytes/leukocytes (%), neutrophils (10^3/mm^3), neutrophils/leukocytes (%), basophils/leukocytes (%), eosinophils (10^3/mm^3), eosinophils/leukocytes (%), monocytes (10^3/mm^3), monocytes/leukocytes (%). Clinical chemistry included parameters: aspartate aminotransferase (units per liter [U/L]) (>3.0* ULN), alanine aminotransferase (U/L) (>3.0* ULN), alkaline phosphatase (U/L) (>3.0* ULN), creatinine (milligram per deciliter [mg/dL]) (>1.3* ULN), potassium (milliequivalent per liter [mEq/L]) (>1.1* ULN), bicarbonate (mEq/L) (>1.1* ULN).
Time Frame: Screening up to Day 29
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
Number analyzed (Participants) | 59 | 58 | 71 | 47
Participants | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to 28 days after last dose of study treatment (maximum up to 60 days)
Description: Same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Safety analysis set included all participants who received at least 1 dose of the investigational product according to actual treatment received.
Arm/Group | Vehicle | Crisaborole Ointment 2% BID | Hydrocortisone Butyrate Cream 0.1% BID | Pimecrolimus Cream 1% BID
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/58 | 0/71 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/58 | 0/71 | 0/47
Other Adverse Events (participants affected / at risk) | 10/59 | 18/58 | 4/71 | 16/47
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle (N=59) | Crisaborole Ointment 2% BID (N=58) | Hydrocortisone Butyrate Cream 0.1% BID (N=71) | Pimecrolimus Cream 1% BID (N=47)
Headache (Nervous system disorders) | 1 | 3 | 2 | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 7 | 4 | 2 | 7
Eczema (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 3 | 0 | 3
Rhinitis (Infections and infestations) | 0 | 2 | 1 | 3
Application site pain (General disorders) | 1 | 8 | 0 | 2

LIMITATIONS AND CAVEATS:
Study was terminated early by sponsor. Decision was not due to safety/efficacy concerns, but was related to business, portfolio reprioritization. Sub-study planned as per Amendment 3 was not initiated, as sub study site setup didn't complete prior to study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/01/NCT03539601/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT03539601/SAP_001.pdf